CLINICAL TRIAL: NCT04977986
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple-Center, Efficacy and Safety Study of ZYN002 Administered as a Transdermal Gel to Children, Adolescents and Young Adults With Fragile X Syndrome - RECONNECT
Brief Title: Clinical Study of Cannabidiol in Children, Adolescents, and Young Adults With Fragile X Syndrome
Acronym: RECONNECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zynerba Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZYN2-CL-033
Record Dates: First submitted 2021-07-20; First posted 2021-07-27 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Fragile X Syndrome
Keywords: Human Genetics and Inherited Disorders; Other human genetics and inherited disorders
MeSH Terms: conditions — Fragile X Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-controlled, multiple center study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo formulated as a clear gel (transdermal delivery)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ZYN002 - transdermal gel (Experimental): Pharmaceutically manufactured. Cannabidiol is formulated as a clear gel for transdermal delivery.
  Interventions: Drug: ZYN002 - transdermal gel
- Placebo transdermal gel (Placebo Comparator): Placebo is formulated as a clear gel for transdermal delivery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZYN002 - transdermal gel — Pharmaceutically manufactured cannabidiol formulated as a clear gel that can be applied to the skin (transdermal delivery)
  Other Names: cannabidiol formulated as a clear gel that can be applied to the skin (transdermal delivery)
  Arms: ZYN002 - transdermal gel
Drug: Placebo — Placebo formulated as a clear gel that can be applied to the skin (transdermal delivery)
  Other Names:
  Placebo Comparator Matching Placebo
  Other Names: Placebo Comparator; Matching Placebo
  Arms: Placebo transdermal gel

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multiple-center study, to assess the efficacy and safety of Cannabidiol administered as ZYN002 for the treatment of children, adolescent, and young adult patients with Fragile X Syndrome (FXS). Eligible participants will participate in up to an 18-week treatment period, where all participants will receive placebo or active study drug. Patients ages 3 to < 30 years will be eligible to participate.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multiple-center study, to assess the efficacy and safety of ZYN002, a pharmaceutically manufactured cannabidiol, formulated as a clear gel that can be applied to the skin (called transdermal delivery), in children, adolescents, and young adults with FXS. 250 male and female patients, ages 3 to < 30 years, will be randomized 1:1 to either trial drug or placebo and will undergo an 18-week treatment period. Randomization will be stratified by gender, methylation status and weight. The study will be comprised of a Screening visit and a combination of seven visits both onsite (face-to-face) and virtual. The assignment of study drug or placebo will be done by a computer-generated system and neither the study doctor, participant or their caregivers will know which treatment is being given to them. The dose of the treatment will depend on the weight of the participants. If the participants weigh less than or equal to 30 kg, they will receive 2 sachets of the gel per day (1 sachet approximately every 12 hours). If the participant weighs more than 30 kg but less than or equal to 50 kg, they will receive 4 sachets of gel per day (2 sachets approximately every 12 hours). Participants who weigh more than 50 kg will receive 6 sachets of gel per day (3 sachets approximately every 12 hours). Parents/ caregivers will be instructed on proper application of the gel. The gel will be applied to clean, dry, intact skin of the upper arms/ shoulders.

Blood samples will be collected for safety analysis of ZYN002. An independent analytical laboratory will also perform CGG repeat and methylation status analyses. Additionally, the parents/caregivers and study doctor will be asked to complete some questionnaires for efficacy and safety assessment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children and adolescents aged 3 to < 30 years, at the time of Screening.
* Patient resides with caregiver who will continue to provide consistent care throughout the study.
* Judged by the Investigator to be in generally good health at Screening based upon the results of medical history, physical exam, 12-lead ECG and clinical laboratory test results. -Laboratory results outside the reference range must be documented as not clinically significant by both the Investigator and Sponsor.
* Participants must have a diagnosis of FXS through molecular documentation of full mutation of the FMR1 gene documented through genetic testing at Screening.
* Patients with a history of seizure disorders must currently be receiving treatment with a stable regimen of no more than two anti-seizure medications (ASMs) for the four weeks preceding study Screening; or must be seizure-free for one year if not currently receiving ASMs.
* Patients taking psychoactive medication(s) should be on a stable regimen of not more than three such medications for at least fours weeks preceding Screening and must maintain that regimen throughout the study. Psychoactive medications include (but are not limited to) antipsychotics, antidepressants, anxiolytics, attention-deficit / hyperactivity disorder (ADHD) medications, and medications for sleep.
* If patients are receiving non-pharmacological, behavioral and/or dietary interventions, they must be stable and have been doing so for three months prior to screening.
* Patients have a body mass index between 12-30 kg/m2 (inclusive) and patients with a body mass index >30 kg/m2 and <40 kg/m2 with normal liver function laboratory values and with no immediate family history of fatty liver disease.
* Females of childbearing potential must have a negative serum pregnancy test at the Screening Visit and a negative serum or urine pregnancy test at all designated visits.
* Patients and parents/caregivers must be adequately informed of the nature and risks of the study and given written informed consent prior to Screening.
* Patients and parents/caregivers agree to abide by all study restrictions and comply with all study procedures, and in the Investigator's opinion, are reliable and willing and able to comply with all protocol requirements and procedures.

Exclusion Criteria:

* Females who are pregnant, nursing or planning a pregnancy; females of childbearing potential and male patients with a partner of childbearing potential who are unwilling or unable to use an acceptable method of contraception as outlined below for the duration of therapy and for three months after the last dose of study medication. Standard acceptable methods of contraception include abstinence (defined as refraining from heterosexual intercourse from screening to three months after the last dose of study medication: abstinence only applicable for females <18 years) or the use of a highly effective method of contraception, including hormonal contraception, diaphragm, cervical cap, vaginal sponge, condom, spermicide, vasectomy, or intrauterine device. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject. Periodic abstinence (calendar, symptothermal, post-ovulation methods) is not an acceptable method of contraception.
* Patient has transitioned to independent living or living in a residential facility such as a university setting or congregate care.
* History of significant allergic condition, significant drug-related hypersensitivity, or allergic reaction to any compound or chemical class related to ZYN002 or its excipients.
* Exposure to any investigational drug or device less than or equal to 30 days prior to Screening or at any time during the study.
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST) or total bilirubin levels greater than or equal to 2 times the upper limit of normal or alkaline phosphatase levels greater than or equal to 3 times the upper limit of normal.
* Use of cannabis or any THC or CBD-containing product within 3 months of Screening Visit or during the study (aside from ZYN002).
* Patient has a positive drug screen, including ethanol, cocaine, THC, barbiturates, amphetamines (unless prescribed), benzodiazepines (except midazolam or comparable administered for blood draws and ECG collection), and opiates.
* Patient is using the following AEDs (medications for the treatment of seizures and/ or epilepsy): clobazam, phenobarbital, ethosuximide, felbamate, carbamazepine, phenytoin, or vigabatrin.
* Patient is using a strong inhibitor/inducer of CYP3A4 or sensitive substrate of CYP3A4 including but not limited to the following medications: midazolam (except single doses administered for the purposes of obtaining blood samples and ECG's), oral ketoconazole, fluconazole, nefazadone, rifampin, alfentanil, alfuzosin, amiodarone, cyclosporine, dasatinib, docetaxol, eplerenone, ergotamine, everolimus, fentanyl, halofantrine, irinotecan, lapatinib, levomethadyl, lumefantrine, nilotinib, pimozide, quinidine, ranolazine, sirolimus, tacrolimus, temsirolimus, toremifene, tretinioin, vincristine, vinorelbine, St. John's Wort, and grapefruit Juice/products.
* Patients may not be taking any benzodiazepines (except single doses administered for the purposes of obtaining blood samples and ECGs) at screening or throughout the study.
* Patient is expected to initiate or change pharmacologic or non-pharmacologic interventions during the course of the study.
* Patient has an advanced, severe, or unstable disease that may interfere with the study outcome evaluations.
* Patient has acute or progressive neurological disease, psychosis, schizophrenia or any other psychiatric disorder or severe mental abnormalities (other than FXS) that are likely to require changes in drug therapy or interfere with the study objectives or ability to adhere to protocol requirements.
* Patient has a positive result for the presence of HBsAg, HCV, or HIV antibodies.
* Patient has known history of cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, cardiac conduction problems, exercise-related cardiac events including syncope and pre-syncope, risk factors for Torsades de pointes (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome), or other serious cardiac problems.
* Any clinically significant condition or abnormal findings at the Screening Visit that would, in the opinion of the Investigator, preclude study participation or interfere with the evaluation of the study medication.
* Any skin disease or condition including eczema, psoriasis, melanoma, acne, contact dermatitis, scarring, imperfections, lesions, tattoos, or discoloration that may affect treatment application, application site assessments or absorption of the trial drug.
* History of treatment for, or evidence of, drug abuse within the past year.
* Previous participation in a ZYN002 study (with the exception of patients who were screen failures in Study ZYN2-CL-016 and did not enter Study ZYN2-CL-017).
* Patient responds "yes" to Question 4 or 5 on the C-SSRS (Children) during Screening or at any time on study.

Ages: 3 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 215 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist-Community Fragile X Factor Structure (ABC-C FXS) Pre-specified Subscale 1 score in patients with complete methylation of the FMR1 gene. | Change from Baseline to Week 18
  The ABC-C FXS is a standard parent/caregiver reported behavioral outcome measure for use in developmental disability clinical trials

SECONDARY OUTCOMES:
Aberrant Behavior Checklist-Community, Fragile X Factor Structure (ABC-C FXS) Pre-specified Subscale 2 in patients with complete methylation of the FMR1 gene. | Change from Baseline to Week 18
  The ABC-C FXS is a standard parent/caregiver reported behavioral outcome measure for use in developmental disability clinical trials
Change on the Caregiver Global Impression of Change (CaGI-C) for Pre-specified parameter among patients with complete methylation of the FMR1 gene. | Change from Baseline to Week 18
  The CaGI-C global impression of change is a 7-point Likert scale designed to measure behavioral symptomatic change at a specific time compared to baseline.
Clinical Global Impression- Improvement (CGI-I) scale among patients with complete methylation of the FMR1 gene. | Change from Baseline to Week 18
  The CGI-I global improvement item is a 7-point Likert scale to rate the behavioral change in a child at a specified time compared to baseline.
Change in ABC-C FXS pre-specified Subscale 1 among all randomized patients (complete and partial methylation of the FMR1 gene). | Change from Baseline to Week 18
  The ABC-C FXS is a standard parent/caregiver reported behavioral outcome measure for use in developmental disability clinical trials
Number of patients with adverse events | Day 1, Week 2, Week 4, Week 6, Week 10, Week 14, Week 18 and through 4-week post-dose telephone follow-up
  Collection of adverse events
Number of participants with abnormal physical and neurological exams | Screening, Day 1 and Week 18
  Physical and neurological exams
Number of participants with abnormal clinical laboratory results | Screening, Week 10 and Week 18
  Laboratory tests and urinalysis
Number of participants with abnormal vital sign results | Screening, Day 1, Week 2 and Week 18
  Vital sign measurements (blood pressure, heart rate, respiratory rate and temperature)
Number of participants with abnormal ECG | Screening and Week 18
  12-lead ECG
Withdrawal characteristics of ZYN002 using the Penn Physician Withdrawal Checklist | Week 18 and 4-week post last dose
  Penn Physician Withdrawal Checklist
Skin tolerability as assessed using daily skin diary | Daily from Day 1 through Week 18
  Daily skin irritation diary

CONTACTS AND LOCATIONS:
Locations (27):
- United States (18):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Science 37, Culver City, California
  - Amnova Clinical Research, LLC, Irvine, California
  - Thompson Autism Center CHOC, Orange, California
  - UC Davis Health System, MIND Institute, Sacramento, California
  - Children's National Medical center, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Rare Disease Research, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Minnesota Fragile X Clinic (Voyager Clinic), Minneapolis, Minnesota
  - University of Mississippi, Jackson, Mississippi
  - The Fragile X Spectrum Disorder Clinic at Icahn School of Medicine at Mount Sinai, Division of Medical Genetics, New York, New York
  - Central States Research, Tulsa, Oklahoma
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Greenwood Genetic Center, Greenville, South Carolina
  - Primary Children's Hospital, Salt Lake City, Utah
- Australia (3):
  - Westmead Children's Hospital, Sydney, New South Wales
  - Lady Cilento Children's Hospital - South Brisbane, Brisbane, Queensland
  - Genetics Clinics Australia, Melbourne, Victoria
- Wellcome HRB Clinical Research Facility, Dublin, Ireland
- Health New Zealand - Te Whatu Ora - Wellington Hospital, Newtown, Wellington Region, New Zealand
- United Kingdom (4):
  - University of Edinburgh, Edinburgh
  - Leicester Clinical Research, Leicester
  - King's College, London
  - Manchester University NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No